CLINICAL TRIAL: NCT02226575
Title: Study of Management and Coaching in Atrial Fibrillation
Brief Title: Management and Coaching in Atrial Fibrillation
Acronym: MANCAF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Helena Ekblad (Other Government)
Collaborators: School of Health Sciences, Jönköping University, Jönköping Sweden (Unknown)
Responsible Party: Sponsor-Investigator, Helena Ekblad, RN, BSC, PhD-student, Region Jönköping County
Organization: Region Jönköping County (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: SMAC-PAFHM11
Record Dates: First submitted 2014-08-19; First posted 2014-08-27 (Estimated); Last update posted 2015-03-06 (Estimated); Status verified 2015-03

CONDITIONS: Atrial Fibrillation
Keywords: Sense of coherence
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Distress management (Experimental): The distress management program (cognitive behavioral therapy) alongside standard care
  Interventions: Behavioral: A cognitive behavior therapy distress management program targeting wellbeing in patients with atrial fibrillation and their relatives
- Control (No Intervention): Controls only dilivery standard care

INTERVENTIONS:
Behavioral: A cognitive behavior therapy distress management program targeting wellbeing in patients with atrial fibrillation and their relatives — Controls only delivery standard care. Experimental group deliver standard care plus a distress management program (cognitive behavioral therapy) performed in groups by a nurse, a pedagogue and a cardiologist (all trained in the distress management program).
  Arms: Distress management

SUMMARY:
The purpose of this study is to evaluate the effect of a cognitive behavior therapy distress management program targeting wellbeing in patients with atrial fibrillation and their relatives.

DETAILED DESCRIPTION:
A randomized controlled design with pre- and 12 month posttest including persons living with atrial fibrillation and their relatives.

The distress management program (cognitive behavioral therapy) delivered in groups by a specialistnurse, a pedagogue and a cardiologist all trained in the distress management program. The program delivered to participants into three group- sessions extensive two hours each during a five weeks period 2011-2013.

Eligible participants were all consecutive identified when discharge after hospital care due to atrial fibrillation. The random process were managed by an open-label computer as block - randomization. Participants were enrolled and randomized during 2011-2013 into two arms; either to an experiment group to the distress management program or the control group. The trial, run alongside the standard care all of the participants received at a cardiology unit in a county hospital. The standard care was required to following actual guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with atrial fibrillation.
* Relative to patient with atrial fibrillation.
* To be over 18 years old .

Exclusion Criteria:

* Unwillingness to participate in the study.
* Other complicating illness'.
* Language difficulties that prevent answering surveys.
* Participation in another study.
* Accommodation outside the hospital's catchment area.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2011-09; Primary Completion 2014-11 (Actual); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in self-rated sense of coherence (13-item); The sense of coherens scale, SOC 13-item at week 52. | baseline and after 12 months
Changes from baseline in self-rated Health related quality of Life (36 item); The SF 36 - item short-form health status survey at week 52 | baseline and after 12 mounth
Changes from baseline in self-rated mastering (7 item); The 7-item Mastery scale at week 52 | baseline and after 12 months

SECONDARY OUTCOMES:
Changes from baseline in self-rated Health related quality of life (5 item); EuroQol Five Dimensions, EQ-5D at week 52 | baseline and after 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Bengt Fridlund, Professor, Principal Investigator — School of Health Sciences, Jönköping University, Jönköping Sweden
Locations (1):
- County Hospital Ryhov, Jönköping, Jönköping County, Sweden

REFERENCES:
- [Background] Thrall G, Lip GY, Carroll D, Lane D. Depression, anxiety, and quality of life in patients with atrial fibrillation. Chest. 2007 Oct;132(4):1259-64. doi: 10.1378/chest.07-0036. Epub 2007 Jul 23. PMID 17646231
- [Background] Dalteg T, Benzein E, Sandgren A, Fridlund B, Malm D. Managing uncertainty in couples living with atrial fibrillation. J Cardiovasc Nurs. 2014 May-Jun;29(3):E1-10. doi: 10.1097/JCN.0b013e3182a180da. PMID 24108265
- [Background] Ekblad H, Ronning H, Fridlund B, Malm D. Patients' well-being: experience and actions in their preventing and handling of atrial fibrillation. Eur J Cardiovasc Nurs. 2013 Apr;12(2):132-9. doi: 10.1177/1474515112457132. Epub 2012 Aug 30. PMID 22936792
- [Background] Lane DA, Langman CM, Lip GY, Nouwen A. Illness perceptions, affective response, and health-related quality of life in patients with atrial fibrillation. J Psychosom Res. 2009 Mar;66(3):203-10. doi: 10.1016/j.jpsychores.2008.10.007. PMID 19232232
- [Background] Kupper N, van den Broek KC, Widdershoven J, Denollet J. Subjectively reported symptoms in patients with persistent atrial fibrillation and emotional distress. Front Psychol. 2013 Apr 24;4:192. doi: 10.3389/fpsyg.2013.00192. eCollection 2013. PMID 23630509
- [Background] Smith D, Lip GY, Lane DA. Impact of symptom control on health-related quality of life in atrial fibrillation patients: the psychologist's viewpoint. Europace. 2010 May;12(5):608-10. doi: 10.1093/europace/euq083. Epub 2010 Mar 30. No abstract available. PMID 20353966
- [Background] Gulliksson M, Burell G, Vessby B, Lundin L, Toss H, Svardsudd K. Randomized controlled trial of cognitive behavioral therapy vs standard treatment to prevent recurrent cardiovascular events in patients with coronary heart disease: Secondary Prevention in Uppsala Primary Health Care project (SUPRIM). Arch Intern Med. 2011 Jan 24;171(2):134-40. doi: 10.1001/archinternmed.2010.510. PMID 21263103
- [Background] Eriksson M, Lindstrom B. Antonovsky's sense of coherence scale and the relation with health: a systematic review. J Epidemiol Community Health. 2006 May;60(5):376-81. doi: 10.1136/jech.2005.041616. PMID 16614325
- [Background] McCabe PJ. Psychological distress in patients diagnosed with atrial fibrillation: the state of the science. J Cardiovasc Nurs. 2010 Jan-Feb;25(1):40-51. doi: 10.1097/JCN.0b013e3181b7be36. PMID 19935428
- [Background] Fjorback LO, Arendt M, Ornbol E, Fink P, Walach H. Mindfulness-based stress reduction and mindfulness-based cognitive therapy: a systematic review of randomized controlled trials. Acta Psychiatr Scand. 2011 Aug;124(2):102-19. doi: 10.1111/j.1600-0447.2011.01704.x. Epub 2011 Apr 28. PMID 21534932
- [Derived] Malm D, Fridlund B, Ekblad H, Karlstrom P, Hag E, Pakpour AH. Effects of brief mindfulness-based cognitive behavioural therapy on health-related quality of life and sense of coherence in atrial fibrillation patients. Eur J Cardiovasc Nurs. 2018 Oct;17(7):589-597. doi: 10.1177/1474515118762796. Epub 2018 Mar 1. PMID 29493266